CLINICAL TRIAL: NCT07314489
Title: A Prospective Cohort Study on the Changes of Glucose Metabolism and Exocrine Function in Patients With Chronic Pancreatitis Complicated With Exocrine Dysfunction After Pancreatic Enzyme Intervention
Brief Title: A Study on the Changes of Glucose Metabolism and Exocrine Function in Patients With Chronic Pancreatitis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025SL054
Record Dates: First submitted 2025-07-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis Pancreatic Exocrine Insufficiency Blood Glucose
Keywords: chronic pancreatitis; pancreatitis; exocrine insufficiency; blood glucose
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Creon（Pancreatin Enteric-coated Capsules） (Active Comparator): For newly diagnosed patients with chronic pancreatitis combined with exocrine insufficiency, administer the Creon capsules and take them regularly for 3 months.
  Interventions: Drug: Creon（Pancreatin Enteric-coated Capsules）

INTERVENTIONS:
Drug: Creon（Pancreatin Enteric-coated Capsules） — This product is a mixture of various enzymes extracted from pig pancreas, mainly including trypsin, pancreatic lipase and pancreatic amylase.Take 1 tablet (0.3g) during meals, 3 times a day.0.3 grams is equivalent to 20,000 European Pharmacopoeia units of pancreatic lipase, 16,000 European Pharmacopoeia units of pancreatic amylase, and 1,200 European Pharmacopoeia units of pancreatic protease.

SUMMARY:
This study aims to investigate the impact of pancreatic exocrine insufficiency on the glucose profile and pancreatic and gastrointestinal endocrine hormones in patients with chronic pancreatitis through pancreatic enzyme intervention in a reverse manner.

The primary objective is to observe the changes in glucose profile following pancreatic enzyme intervention in patients with chronic pancreatitis complicated by exocrine insufficiency and normal glucose metabolism.

The secondary objective is to observe the changes in pancreatic endocrine and exocrine functions and gastrointestinal endocrine hormone levels following pancreatic enzyme intervention in patients with chronic pancreatitis complicated by exocrine insufficiency and normal glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female Chinese subjects aged 18 years or older; 2. Patients with a clear diagnosis of chronic pancreatitis; 3. Glycated hemoglobin (HbA1c) levels between 4% and 6%; 4. FE-1 < 100 µg/g.

Exclusion Criteria:

* 1. A history of diabetes or prediabetes, or preoperative glycated hemoglobin (HbA1c) ≥ 6.0% or fasting venous glucose ≥ 6.1 mmol/L; 2. Positive for islet-related antibodies; 3. Patients who are currently receiving or have previously received pancreatic enzyme replacement therapy (PERT); 4. Allergy to the components of PERT drugs; 5. Exocrine pancreatic insufficiency (EPI) caused by other reasons, such as post-gastrectomy or post-intestinal resection; 6. Undergoing pancreatic surgery other than endoscopic retrograde cholangiopancreatography (ERCP); 7. Renal disease of stage G3, G4, or G5; 8. Decompensated chronic liver disease; 9. Receiving glucocorticoid therapy; 10. Pregnant or breastfeeding women; 11. Patients with malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in glucose profile before and after pancreatic enzyme intervention | From enrollment to 3 months after pancreatic enzyme intervention

SECONDARY OUTCOMES:
Measure the changes in pancreatic endocrine and exocrine functions and gastrointestinal endocrine hormone levels after pancreatic enzyme intervention. | From enrollment to 3 months after pancreatic enzyme intervention

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Changzheng Hospital, Shanghai